CLINICAL TRIAL: NCT03348514
Title: A Phase 1, First-in-Human, Safety, Dose Tolerance, Pharmacokinetics, and Pharmacodynamics Study of CPX-POM in Patients With Advanced Solid Tumors.
Brief Title: Safety, Dose Tolerance, Pharmacokinetics, and Pharmacodynamics Study of CPX-POM in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CicloMed LLC (Industry)
Collaborators: Cmed Clinical Services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CPX-POM-01-001
Record Dates: First submitted 2017-11-15; First posted 2017-11-21 (Actual); Results first posted 2021-11-17 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: This is a Phase I, first-in-human, multicenter, open label, dose escalating study to evaluate the DLTs and MTD and to determine the recommended Phase 2 dose (RP2D) of CPX-POM administered IV in patients with any histologically- or cytologically-confirmed solid tumor type.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- CPX-POM - 30 mg/m^2 (Experimental)
  Interventions: Drug: CPX-POM - 30 mg/m^2
- CPX-POM - 60 mg/m^2 (Experimental)
  Interventions: Drug: CPX-POM - 60 mg/m^2
- CPX-POM - 120 mg/m^2 (Experimental)
  Interventions: Drug: CPX-POM - 120 mg/m^2
- CPX-POM - 240 mg/m^2 (Experimental)
  Interventions: Drug: CPX-POM - 240 mg/m^2
- CPX-POM - 360 mg/m^2 (Experimental)
  Interventions: Drug: CPX-POM - 360 mg/m^2
- CPX-POM - 600 mg/m^2 (Experimental)
  Interventions: Drug: CPX-POM - 600 mg/m^2
- CPX-POM - 900 mg/m^2 (Experimental)
  Interventions: Drug: CPX-POM - 900 mg/m^2
- CPX-POM - 1200 mg/m^2 (Experimental)
  Interventions: Drug: CPX-POM - 1200 mg/m^2

INTERVENTIONS:
Drug: CPX-POM - 30 mg/m^2 — CPX-POM
  Arms: CPX-POM - 30 mg/m^2
Drug: CPX-POM - 60 mg/m^2 — CPX-POM
  Arms: CPX-POM - 60 mg/m^2
Drug: CPX-POM - 120 mg/m^2 — CPX-POM
  Arms: CPX-POM - 120 mg/m^2
Drug: CPX-POM - 240 mg/m^2 — CPX-POM
  Arms: CPX-POM - 240 mg/m^2
Drug: CPX-POM - 360 mg/m^2 — CPX-POM
  Arms: CPX-POM - 360 mg/m^2
Drug: CPX-POM - 600 mg/m^2 — CPX-POM
  Arms: CPX-POM - 600 mg/m^2
Drug: CPX-POM - 900 mg/m^2 — CPX-POM
  Arms: CPX-POM - 900 mg/m^2
Drug: CPX-POM - 1200 mg/m^2 — CPX-POM
  Arms: CPX-POM - 1200 mg/m^2

SUMMARY:
This is a first-in-human, Phase I, multicenter, open label, dose escalation study to evaluate the DLTs and MTD and to determine the recommended Phase 2 dose (RP2D) of CPX-POM administered IV in patients with any histologically- or cytologically-confirmed solid tumor type.

DETAILED DESCRIPTION:
The study will initially employ an accelerated escalation design, with a single patient enrolled in each cohort (i.e., Single-Patient Cohorts). The initial patient will receive CPX-POM at a starting dose of 30 mg/m2. Doses will be escalated (doubling), until a ≥Grade 2 toxicity (with the exception of alopecia), is encountered. Subsequently that and all subsequent cohorts will follow a classical "3+3" dose escalation design.

Note: Fosciclopirox is the generic name for CPX-POM.

ELIGIBILITY:
Inclusion Criteria Include:

1. Patient is male or female aged ≥18 years.
2. Patient provided signed and dated informed consent prior to initiation of any study procedures.
3. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 (fully active, able to carry out all pre-disease activities without restriction) or 1 (unable to perform physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature).
4. Patient has a predicted life expectancy of ≥3 months.
5. Dose escalation cohorts only: Patient has adequate renal function (creatinine ≤1.5 × the upper limit of normal [ULN]) or a glomerular filtration rate (GFR) of ≥50 mL/min/1.73 m^2). Expansion cohort only: Patient has a GFR of ≥30 mL/min/1.73 m^2.
6. Patient has adequate hepatic function, as evidenced by a total bilirubin ≤1.5 × ULN, aspartate transaminase (AST), and /or alanine transaminase (ALT) ≤3 × ULN or ≤5 ×ULN, if due to liver involvement by tumor.
7. Patient has adequate bone marrow function, as evidenced by hemoglobin ≥9.0 g/dL in the absence of transfusion within the previous 72 hours, platelet count ≥100×10^9cells/L, and absolute neutrophil count (ANC) ≥1.5×10^9 cells/L.
8. Patient has no significant ischemic heart disease or myocardial infarction (MI) within 6 months before the first dose of CPX-POM and currently has adequate cardiac function, as evidenced by a left ventricular ejection fraction of >50% as assessed by multi-gated acquisition (MUGA) or ultrasound/echocardiography (ECHO); and corrected QT interval (QTc) <470 msec by Fridericia (QTcF). The eligibility of patients with ventricular pacemakers for whom the QT interval may not be accurately measurable will be determined on a case-by-case basis by the Sponsor in consultation with the Medical Monitor.
9. Patient and his/her partner agree to use adequate contraception after providing written informed consent through 3 months after the last dose of CPX-POM, as follows:

   1. For women: Negative pregnancy test during Screening and at Day 1 of each treatment cycle and compliant with a medically-approved contraceptive regimen during and for 3 months after the treatment period or documented to be surgically sterile or postmenopausal.
   2. For men: Compliant with a medically-approved contraceptive regimen during and for 3 months after the treatment period or documented to be surgically sterile. Men whose sexual partners are of child-bearing potential must agree to use 2 methods of contraception prior to study entry, during the study, and for 3 months after the treatment period.
10. Patient is willing and able to participate in the study and comply with all study requirements.

Exclusion Criteria Include:

Patients who meet any of the following exclusion criteria are not to be enrolled in this study

1. Patient has a history of risk factors for torsade de pointes (e.g., heart failure, hypokalemia, family history of long QT syndrome) or requires the use of concomitant medications that prolong the QT/QTc interval during study participation. Patients should not receive anti-emetic medications before and following Dose 1 of Cycle 1 for each treatment cohort. However, anti-emetics such as ondansetron or granisetron that have a mild QTc prolonging effect are allowed starting with Dose 2 of Cycle 1, if used with caution and attention to the approved labelling.
2. Patient has an abnormal cardiac appearance/heart size, as evidenced by chest X-ray or computed tomography (CT) scan.
3. Patient has an uncontrolled or severe intercurrent medical condition (including uncontrolled brain metastases). Patients with stable brain metastases either treated or being treated with a stable dose of steroids/anticonvulsants, with no dose change within 4 weeks before the first dose of CPX-POM and no anticipated dose change, are allowed. The decision to exclude a patient from the study for an uncontrolled or severe intercurrent medical condition will be made by the Principal Investigator. Examples could include epilepsy, resistant infection, or any other neurological disease that would make clinical assessment difficult.
4. Patient underwent major surgery within 4 weeks before the first dose of CPX-POM or received cancer-directed therapy (chemotherapy, radiotherapy, hormonal therapy, biologic or immunotherapy, etc.) or an drug or device within 4 weeks (6 weeks for mitomycin C and nitrosoureas) or 5 half-lives of that agent (whichever is shorter) before the first dose of CPX-POM. A minimum of 10 days between termination of the investigational drug and administration of CPX-POM is required. In addition, any drug-related toxicity, with the exception of alopecia, should have recovered to ≤Grade 1.
5. If female, patient is pregnant or breast-feeding.
6. Patient has evidence of a serious active infection (e.g., infection requiring treatment with intravenous antibiotics).
7. Patient has active Hepatitis A infection.
8. Patient known human immunodeficiency virus (HIV) or Hepatitis B or C infection, as such patients may be at increased risk for toxicity due to concomitant treatment and disease-related symptoms may preclude accurate assessment of the safety of CPX POM.
9. Patient has an important medical illness or abnormal laboratory finding that, in the Investigator's opinion, would increase the risk of participating in this study.
10. Patient is taking warfarin.
11. Patient has a history of other malignancy treated with curative intent within the previous 5 years with the exception of adequately treated non-melanoma skin cancer or carcinoma in situ of the cervix. Patients with previous invasive cancers are eligible if the treatment was completed more than 5 years prior to initiating current study treatment, and there is no evidence of recurrent disease.
12. Patient has known allergy or hypersensitivity to components of CPX-POM.
13. Patient is taking any iron replacement therapy administered IV, IM, or orally due to the potential for loss of anticancer activity due to drug and metabolites chelating iron.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Taylor III, MD, MSc, Principal Investigator — University of Kansas Medical Center
Locations (5):
- United States (5):
  - Sarah Cannon Research Institute, Denver, Colorado
  - Florida Cancer Specialists & Research Institute, Sarasota, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Tennessee Oncology PLLC, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Weir SJ, Dandawate P, Standing D, Bhattacharyya S, Ramamoorthy P, Rangarajan P, Wood R, Brinker AE, Woolbright BL, Tanol M, Ham T, McCulloch W, Dalton M, Reed GA, Baltezor MJ, Jensen RA, Taylor JA 3rd, Anant S. Fosciclopirox suppresses growth of high-grade urothelial cancer by targeting the gamma-secretase complex. Cell Death Dis. 2021 May 31;12(6):562. doi: 10.1038/s41419-021-03836-z. PMID 34059639
- [Derived] Weir SJ, Wood R, Schorno K, Brinker AE, Ramamoorthy P, Heppert K, Rajewski L, Tanol M, Ham T, McKenna MJ, McCulloch W, Dalton M, Reed GA, Jensen RA, Baltezor MJ, Anant S, Taylor JA 3rd. Preclinical Pharmacokinetics of Fosciclopirox, a Novel Treatment of Urothelial Cancers, in Rats and Dogs. J Pharmacol Exp Ther. 2019 Aug;370(2):148-159. doi: 10.1124/jpet.119.257972. Epub 2019 May 21. PMID 31113837

RESULTS

PARTICIPANT FLOW:
Groups:
- CPX-POM - 30 mg/m^2: Period 1, Dose Cohort - 30 mg/m^2
- CPX-POM - 60 mg/m^2: Period 2, Dose Cohort - 60 mg/m^2
- CPX-POM - 120 mg/m^2: Period 3, Dose Cohort - 120 mg/m^2
- CPX-POM - 240 mg/m^2: Period 4, Dose Cohort - 240 mg/m^2
- CPX-POM - 360 mg/m^2: Period 5, Dose Cohort - 360 mg/m^2
- CPX-POM - 600 mg/m^2: Period 6, Dose Cohort - 600 mg/m^2
- CPX-POM - 900 mg/m^2: Period 7, Dose Cohort - 900 mg/m^2
- CPX-POM - 1200 mg/m^2: Period 8, Dose Cohort - 1200 mg/m^2
Period: Overall Study
Arm/Group | CPX-POM - 30 mg/m^2 | CPX-POM - 60 mg/m^2 | CPX-POM - 120 mg/m^2 | CPX-POM - 240 mg/m^2 | CPX-POM - 360 mg/m^2 | CPX-POM - 600 mg/m^2 | CPX-POM - 900 mg/m^2 | CPX-POM - 1200 mg/m^2
Started | 1 | 1 | 1 | 1 | 3 | 4 | 6 | 2
Completed | 1 | 1 | 1 | 1 | 3 | 4 | 6 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- CPX-POM - 30 mg/m^2: Period1, Dose Cohort - 30 mg/m^2
- Total: Total of all reporting groups
Arm/Group | CPX-POM - 30 mg/m^2 | CPX-POM - 60 mg/m^2 | CPX-POM - 120 mg/m^2 | CPX-POM - 240 mg/m^2 | CPX-POM - 360 mg/m^2 | CPX-POM - 600 mg/m^2 | CPX-POM - 900 mg/m^2 | CPX-POM - 1200 mg/m^2 | Total
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 4 | 6 | 2 | 19
Age, Continuous [Mean (Full Range); unit: years] | 46 | 62 | 76 | 61 | 54 [20 to 82] | 63 [57 to 72] | 60 [38 to 70] | 82.5 [79 to 86] | 63 [20 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 1 | 2 | 4 | 4 | 0 | 13
  Male | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 1 | 1 | 1 | 1 | 3 | 4 | 5 | 2 | 18
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cancer type [Count of Participants; unit: Participants]
  Colon | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 5
  Bladder | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Breast | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Gastric | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Head and Neck | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Liver | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Ovarian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Prostate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Other | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) of CPX-POM
Description: The primary objective of this study is to evaluate the dose limiting toxicities (DLTs) of ciclopirox phosphoryloxymethyl ester (CPX-POM) administered intravenously (IV) and establish the CPX POM dose recommended for further investigation.
  A DLT will include some Grade 3 or 4 AEs (as assessed by CTCAE version 4.03) if deemed related to study drug. In addition, any patient who is unable to receive 80% of the expected dose of CPX-POM (i.e., patients who are unable to receive at least 4 of the 5 scheduled doses) because of AEs will be considered to have a DLT.
  In order to identify any DLTs, safety assessments including AEs, physical examinations, vital signs, and clinical laboratory tests will be conducted during each study visit through Day 22.
Time Frame: Up to 22 days for each cohort
Measure: Number; unit: participants
Arm/Group | CPX-POM - 30 mg/m^2 | CPX-POM - 60 mg/m^2 | CPX-POM - 120 mg/m^2 | CPX-POM - 240 mg/m^2 | CPX-POM - 360 mg/m^2 | CPX-POM - 600 mg/m^2 | CPX-POM - 900 mg/m^2 | CPX-POM - 1200 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 4 | 6 | 2
participants
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Grade 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0

2. Primary Outcome: Determine the Maximum Tolerated Dose (MTD) of CPX-POM
Description: The primary objective of this study is to evaluate the maximum tolerated dose (MTD) of ciclopirox phosphoryloxymethyl ester (CPX-POM) administered intravenously (IV) and establish the CPX POM dose recommended for further investigation. MTD was determined by testing increasing doses up to 1200 mg/m^2 by IV.
  The MTD is defined as the dose BELOW that dose which causes DLTs in ≥33% of patients.
Time Frame: Days 1, 2, 3, 4, 5, 6, 10, 22 and 28
Measure: Number; unit: mg/m^2
Groups:
- All Participants: All participants who received at least one dose of CPX-POM either at 30 mg/m^2, 60 mg/m^2, 120 mg/m^2, 240 mg/m^2, 360 mg/m^2, 600 mg/m^2, 900 mg/m^2 and 1200 mg/m^2 via IV.
Arm/Group | All Participants
Number analyzed (Participants) | 19
mg/m^2 | 900

3. Secondary Outcome: Assess Plasma PK: Cmax (ng/mL) of the Active Metabolite, Ciclopirox (CPX), Following Five Consecutive Days of Once Daily Dosing.
Description: Measure PK parameter Cmax (ng/mL)
Time Frame: Days 5-6
Population: Pharmacokinetic data not obtained in one patient receiving 1200 mg/m^2
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- CPX-POM - 120 mg/m^2: Period 3, Cohort Dose - 120 mg/m^2
- CPX-POM - 240 mg/m^2: Period 4, Cohort Dose - 240 mg/m^2
Arm/Group | CPX-POM - 30 mg/m^2 | CPX-POM - 60 mg/m^2 | CPX-POM - 120 mg/m^2 | CPX-POM - 240 mg/m^2 | CPX-POM - 360 mg/m^2 | CPX-POM - 600 mg/m^2 | CPX-POM - 900 mg/m^2 | CPX-POM - 1200 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 4 | 6 | 1
ng/mL | 371 | 1935 | 3491 | 6792 | 5297 (1182) | 9457 (512) | 17277 (1913) | 15970

4. Secondary Outcome: Assess Plasma PK: Terminal Half-life of the Active Metabolite, Ciclopirox (CPX), Following Five Consecutive Days of Once Daily Dosing.
Description: Determine Terminal Half-Life
Time Frame: Days 5-6
Population: Pharmacokinetic data not obtained in one patient receiving 1200 mg/m^2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | CPX-POM - 30 mg/m^2 | CPX-POM - 60 mg/m^2 | CPX-POM - 120 mg/m^2 | CPX-POM - 240 mg/m^2 | CPX-POM - 360 mg/m^2 | CPX-POM - 600 mg/m^2 | CPX-POM - 900 mg/m^2 | CPX-POM - 1200 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 4 | 6 | 1
hours | 2.34 | 0.54 | 5.56 | 3.34 | 3.12 (1.34) | 4.61 (1.46) | 8.30 (2.63) | 7.43

5. Secondary Outcome: Assess Plasma PK: AUCss (ng/mL/hr) of the Active Metabolite, Ciclopirox (CPX), Following Five Consecutive Days of Once Daily Dosing.
Description: Measure PK parameter area-under-the-plasma-drug/metabolite-concentration-time curve (ng/mL/hr) following single dose (AUC) and at steady-state AUCss following single and repeat drug administration.
Time Frame: Days 5-6
Population: Pharmacokinetic data not obtained in one patient receiving 1200 mg/m^2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | CPX-POM - 30 mg/m^2 | CPX-POM - 60 mg/m^2 | CPX-POM - 120 mg/m^2 | CPX-POM - 240 mg/m^2 | CPX-POM - 360 mg/m^2 | CPX-POM - 600 mg/m^2 | CPX-POM - 900 mg/m^2 | CPX-POM - 1200 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 4 | 6 | 1
ng*hr/mL
  Single Dose AUCs | 589 | 1262 | 3736 | 4622 | 4731 (1310) | 11914 (1852) | 24148 (6067) | 34470
  Steady State AUCss | 515 | 1328 | 5143 | 6000 | 4856 (910) | 12484 (1182) | 23414 (1913) | 28048

6. Secondary Outcome: Assess Plasma PK: Cls (mL/hr/kg) of the Active Metabolite, Ciclopirox (CPX), Following Five Consecutive Days of Once Daily Dosing.
Description: Measure PK parameter Cls (mL/hr/kg) - systemic clearance following single dose (Cls) following single and repeat drug administration.
Time Frame: Days 5-6
Population: Pharmacokinetic data not obtained in one patient receiving 1200 mg/m^2
Measure: Mean (Standard Deviation); unit: mL/hr/kg
Arm/Group | CPX-POM - 30 mg/m^2 | CPX-POM - 60 mg/m^2 | CPX-POM - 120 mg/m^2 | CPX-POM - 240 mg/m^2 | CPX-POM - 360 mg/m^2 | CPX-POM - 600 mg/m^2 | CPX-POM - 900 mg/m^2 | CPX-POM - 1200 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 4 | 6 | 1
mL/hr/kg
  Single Dose Cls | 614 | 581 | 361 | 515 | 1065 (435) | 507 (95) | 432 (142) | 375
  Steady State Cls | 702 | 552 | 262 | 397 | 963 (271) | 471 (113) | 421 (184) | 456

7. Secondary Outcome: Assess Plasma PK: Vd and Vss (mL/kg) of the Active Metabolite, Ciclopirox (CPX), Following Five Consecutive Days of Once Daily Dosing.
Description: Measure PK parameters Vd (apparent volume of distribution) and Vss (steady state volume of distribution) (mL/kg)
Time Frame: Days 5-6
Population: Pharmacokinetic data not obtained in one patient receiving 1200 mg/m^2
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | CPX-POM - 30 mg/m^2 | CPX-POM - 60 mg/m^2 | CPX-POM - 120 mg/m^2 | CPX-POM - 240 mg/m^2 | CPX-POM - 360 mg/m^2 | CPX-POM - 600 mg/m^2 | CPX-POM - 900 mg/m^2 | CPX-POM - 1200 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 4 | 6 | 1
mL/kg
  Vd | 2370 | 429 | 2100 | 1966 | 4522 (2715) | 3090 (1015) | 5340 (3935) | 4887
  Vss | 2053 | 473 | 1633 | 736 | 1986 (802) | 1346 (349) | 2261 (1249) | 2518

8. Secondary Outcome: Characterize Plasma PK: AUCss/AUCi Accumulation Ratio of the Active Metabolite, Ciclopirox (CPX), Following Five Consecutive Days of Once Daily Dosing.
Description: Determine PK parameter AUC derived accumulation ratio (AUCss/AUCi ratio)
Time Frame: Days 5-6
Population: Pharmacokinetic data not obtained in one patient receiving 1200 mg/m^2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | CPX-POM - 30 mg/m^2 | CPX-POM - 60 mg/m^2 | CPX-POM - 120 mg/m^2 | CPX-POM - 240 mg/m^2 | CPX-POM - 360 mg/m^2 | CPX-POM - 600 mg/m^2 | CPX-POM - 900 mg/m^2 | CPX-POM - 1200 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 4 | 6 | 1
ratio | 0.86 | 1.05 | 1.59 | 1.30 | 1.08 (0.14) | 1.09 (0.17) | 1.03 (0.29) | 0.81

9. Secondary Outcome: Assess Urine PK: Percent (%) of the CPX-POM Dose Excreted in Urine as CPX-POM and Metabolites, Following Five Consecutive Days of Once Daily Dosing.
Description: Measure Percent Dose (%)
Time Frame: Days 5-6
Population: Urine pharmacokinetic data not obtained in one patient receiving 600 mg/m^2 and one patient receiving 1200 mg/m^2
Measure: Mean (Standard Deviation); unit: Percent of CPX-POM dose
Arm/Group | CPX-POM - 30 mg/m^2 | CPX-POM - 60 mg/m^2 | CPX-POM - 120 mg/m^2 | CPX-POM - 240 mg/m^2 | CPX-POM - 360 mg/m^2 | CPX-POM - 600 mg/m^2 | CPX-POM - 900 mg/m^2 | CPX-POM - 1200 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 3 | 6 | 1
Percent of CPX-POM dose
  % CPX-POM Dose Excreted as CPX-POM over 24 hours | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  % CPX-POM Dose Excreted as ciclopirox over 24 hours | 0.81 | 0.82 | 1.74 | 1.25 | 0.80 (0.21) | 1.21 (0.11) | 4.42 (4.68) | 2.89
  % CPX-POM Dose Excreted as ciclopirox glucuronide over 24 hours | 59.74 | 69.73 | 70.21 | 73.86 | 75.99 (10.40) | 50.70 (29.28) | 69.62 (15.16) | 68.19

10. Secondary Outcome: Assess Urine PK: Average 24-hour Urine Concentration of the Active Metabolite, Ciclopirox (CPX), Following Five Consecutive Days of Once Daily Dosing.
Description: Measure urine CPX concentration (uM)
Time Frame: Days 5-6
Population: Urine pharmacokinetic data not obtained in one patient receiving 600 mg/m^2 and one patient receiving 1200 mg/m^2
Measure: Mean (Standard Deviation); unit: uM
Arm/Group | CPX-POM - 30 mg/m^2 | CPX-POM - 60 mg/m^2 | CPX-POM - 120 mg/m^2 | CPX-POM - 240 mg/m^2 | CPX-POM - 360 mg/m^2 | CPX-POM - 600 mg/m^2 | CPX-POM - 900 mg/m^2 | CPX-POM - 1200 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 3 | 6 | 1
uM | 0.65 | 0.84 | 10.77 | 3.93 | 5.10 (0.86) | 22.91 (12.83) | 138.17 (157.97) | 208.65

ADVERSE EVENTS:
Time Frame: 28 days
Groups:
- CPX-POM - 900 mg/m^2: Period 7 Dose Cohort - 900 mg/m^2
Arm/Group | CPX-POM - 30 mg/m^2 | CPX-POM - 60 mg/m^2 | CPX-POM - 120 mg/m^2 | CPX-POM - 240 mg/m^2 | CPX-POM - 360 mg/m^2 | CPX-POM - 600 mg/m^2 | CPX-POM - 900 mg/m^2 | CPX-POM - 1200 mg/m^2
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/1 | 0/1 | 0/1 | 0/3 | 0/4 | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1 | 0/1 | 0/1 | 1/3 | 3/4 | 1/6 | 1/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 1/1 | 1/1 | 1/3 | 3/4 | 6/6 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CPX-POM - 30 mg/m^2 (N=1) | CPX-POM - 60 mg/m^2 (N=1) | CPX-POM - 120 mg/m^2 (N=1) | CPX-POM - 240 mg/m^2 (N=1) | CPX-POM - 360 mg/m^2 (N=3) | CPX-POM - 600 mg/m^2 (N=4) | CPX-POM - 900 mg/m^2 (N=6) | CPX-POM - 1200 mg/m^2 (N=2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CPX-POM - 30 mg/m^2 (N=1) | CPX-POM - 60 mg/m^2 (N=1) | CPX-POM - 120 mg/m^2 (N=1) | CPX-POM - 240 mg/m^2 (N=1) | CPX-POM - 360 mg/m^2 (N=3) | CPX-POM - 600 mg/m^2 (N=4) | CPX-POM - 900 mg/m^2 (N=6) | CPX-POM - 1200 mg/m^2 (N=2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Taste Disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT03348514/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-02): https://cdn.clinicaltrials.gov/large-docs/14/NCT03348514/SAP_001.pdf